CLINICAL TRIAL: NCT06147960
Title: Evaluation of the Prognostic Role of Inhibitor of Apoptosis Protein Overexpression on the 24-month Recurrence Rate in Locally Advanced Cervical Cancer
Brief Title: Prognostic Role of Inhibitor of Apoptosis Protein Overexpression on Recurrence Rate in Cervical Cancer
Acronym: EPIcol
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2023-1/FF-01
Record Dates: First submitted 2023-11-13; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Cancer of Cervix; Apoptosis
Keywords: Apoptosis inhibiting proteins; Cervical cancer; Apoptosis
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Cervical biopsy specimens. Immunohistochemistry: blocks containing formalin-fixed, paraffin-embedded (FFPE) biopsies will be used to analyse the expression of XIAP, cIAP1 and cIAP2 proteins by immunohistochemistry.
  Evaluation of recurrence according to RECIST v1.1 criteria.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Immunohistochemistry — Blocks containing formalin-fixed, paraffin-embedded (FFPE) biopsies will be used to analyse the expression of XIAP, cIAP1 and cIAP2 proteins by immunohistochemistry. The antibodies will be selected on the basis of the literature and their validation for this technology (Schnoell et al. 2020). The immunohistochemical techniques will be performed on an automated immunolabelling machine (DakoLink®) after antigen demasking. The specific binding of primary antibodies will be revealed by the application of Flex reagent (Dako Agilent), a dextran polymer coupled on the one hand to anti-mouse and anti-rabbit immunoglobulins, and on the other hand to a large number of horseradish peroxidase (HRP) molecules. 3,3'-Diaminobenzidine (DAB) will be used as a substrate for this enzyme to highlight the specific expression of the biomarker. The use of an automated system will ensure the reproducibility of inter-sample labelling.

SUMMARY:
Overexpression of inhibitors of apoptosis proteins (IAPs) in patients treated for locally advanced cervical cancer with exclusive radio-chemotherapy may have a prognostic role on the local recurrence rate at 24 months.

DETAILED DESCRIPTION:
Cervical cancer remains one of the most common cancers in women in terms of both incidence and mortality. Human Papilloma Virus carriage is a necessary condition for the development of these cancers but is not the only factor responsible for malignant transformation. Numerous molecular alterations come into play in the development of these tumours, involving the activation of oncogenes or the inactivation of tumour suppressor genes. Treatment of locally-advanced cancer is based on radiotherapy or a combination of radiotherapy and chemotherapy. Responses to anti-neoplastic treatments remain very heterogeneous from one woman to another. Predicting the response to these treatments would make it possible to envisage early therapeutic alternatives for patients identified as not very sensitive to standard treatments. IAPs (inhibitors of apoptosis proteins), which include XIAP, cIAP1 and cIAP2, are proteins involved in many cancers and capable of downregulating tumour cell apoptosis. It seems justified to investigate the role of these IAPs in resisting apoptosis-inducing anti-neoplastic treatments such as chemotherapy or radiotherapy. The aim of our study is to assess the prognostic role of overexpression of IAPs in locally advanced cervical cancer treated exclusively with radio-chemotherapy. This research seems all the more important as IAP-inhibiting molecules are currently being studied in other types of cancer (ear, nose and throat cancers) and appear to have a very encouraging radiosensitising effect. The hypothesis is that overexpression of IAPs in patients treated for locally advanced cervical cancer with exclusive radio-chemotherapy has a prognostic role on the local recurrence rate at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with the exclusive radio-chemotherapy combination for locally advanced cervical carcinoma (stage Ib-IVb according to FIGO classification).
* Patients aged ≥ 18 years.
* Patients with a minimum of 2 years post-treatment follow-up.
* Patients for whom the initial biopsy specimen (before treatment) is available.
* Patients who have not indicated that they do not wish to participate in the study.
* Patients affiliated to or benefiting from a health insurance scheme.

Exclusion Criteria:

* Patients under court protection, guardianship or curatorship.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — All patients with a cervix
Study Population: The study population is made up of women treated with the exclusive radio-chemotherapy combination for locally advanced cervical carcinoma, managed at the Montpellier Institute of Cancer and Montpellier and Nîmes University Hospitals.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Prognostic role of overexpression of XIAP on the rate of local recurrence in patients treated for locally advanced cervical cancer. | Baseline
  Overexpression of the Inhibitor of Apoptosis Proteins XIAP will be measured to evaluate its prognostic role on the rate of local recurrence at 24 months follow-up in patients treated for locally advanced cervical cancer. The H-score for XIAP will be recorded on a scale of 0 to 300 based on the intensity of carcinoma cells.
Prognostic role of overexpression of XIAP on the rate of local recurrence at 24 months follow-up in patients treated for locally advanced cervical cancer. | 24 months
  Overexpression of the Inhibitor of Apoptosis Proteins XIAP will be measured to evaluate its prognostic role on the rate of local recurrence at 24 months follow-up in patients treated for locally advanced cervical cancer. The H-score for XIAP will be recorded on a scale of 0 to 300 based on the intensity of carcinoma cells.
Prognostic role of overexpression of cIAP1 on the rate of local recurrence in patients treated for locally advanced cervical cancer. | Baseline
  Overexpression of Inhibitors of the Apoptosis Protein cIAP1 will be measured to evaluate its prognostic role on the rate of local recurrence at 24 months follow-up in patients treated for locally advanced cervical cancer.The H-score for cIAP1 be recorded on a scale of 0 to 300 based on the intensity of carcinoma cells.
Prognostic role of overexpression of cIAP1 on the rate of local recurrence at 24 months follow-up in patients treated for locally advanced cervical cancer. | 24 months
  Overexpression of the Inhibitor of Apoptosis Protein cIAP1 will be measured to evaluate its prognostic role on the rate of local recurrence at 24 months follow-up in patients treated for locally advanced cervical cancer.The H-score for cIAP1 be recorded on a scale of 0 to 300 based on the intensity of carcinoma cells.
Prognostic role of overexpression of cIAP2 on the rate of local recurrence in patients treated for locally advanced cervical cancer. | Baseline
  Overexpression of the Inhibitor of Apoptosis Protein cIAP2 will be measured to evaluate its prognostic role on the rate of local recurrence at 24 months follow-up in patients treated for locally advanced cervical cancer.The H-score for cIAP2 be recorded on a scale of 0 to 300 based on the intensity of carcinoma cells.
Prognostic role of overexpression of cIAP2 on the rate of local recurrence at 24 months follow-up in patients treated for locally advanced cervical cancer. | 24 months
  Overexpression of the Inhibitor of Apoptosis Protein cIAP2 will be measured to evaluate its prognostic role on the rate of local recurrence at 24 months follow-up in patients treated for locally advanced cervical cancer. The H-score for cIAP1 be recorded on a scale of 0 to 300 based on the intensity of carcinoma cells.
Local recurrence of cervical cancer | Overall survival at 24 months follow-up in patients treated for locally advanced cervical cancer.
  Local recurrence of cervical cancer at 24 months follow-up according to RECIST v1.1 criteria: Yes/No.
  RECIST 1.1 is a standard way to measure the response of a tumor to treatment in which Complete Response = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. Partial Response = At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
A. Overall survival in patients treated for locally advanced cervical cancer at baseline. | Baseline
  Death will be recorded as YES/NO
A. Overall survival at 24 months follow-up in patients treated for locally advanced cervical cancer. | 24 months
  Death will be recorded as YES/NO
B. Progression-free survival in patients treated for locally advanced cervical cancer. | Baseline
  The time from diagnosis to death from any cause will be recorded in months and days.
B. Progression-free survival at 24 months follow-up in patients treated for locally advanced cervical cancer. | 24 months
  The time from diagnosis to death from any cause will be recorded in months and days.
B. Progression-free survival in patients treated for locally advanced cervical cancer: RECIST criteria | Baseline
  The time between diagnosis and progression according to v1.1 of the RECIST criteria or death from any cause will be recorded in days.
  RECIST 1.1 is a standard way to measure the response of a tumor to treatment in which Complete Response = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. Partial Response = At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
B. Progression-free survival at 24 months follow-up in patients treated for locally advanced cervical cancer: RECIST criteria | 24 months
  The time between diagnosis and progression according to v1.1 of the RECIST criteria or death from any cause will be recorded in days.
  RECIST 1.1 is a standard way to measure the response of a tumor to treatment in which Complete Response = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. Partial Response = At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
B. Progression-free survival in patients treated for locally advanced cervical cancer. H-score | Baseline
  The histochemical scoring assessment (H-SCORE) will be recorded on a scale of 0-300
B. Progression-free survival at 24 months follow-up in patients treated for locally advanced cervical cancer: H-score | 24 months
  The histochemical scoring assessment (H-SCORE) will be recorded on a scale of 0-300
C. Correlation between the Inhibitor of Apoptosis Protein XIAP expression and Programmed Death - Ligand 1 expression. | Baseline
  The expression level of XIAP and the expression level of PD-L1 in biopsies will be measured by immunohistochemistry.
C. Correlation between the Inhibitor of Apoptosis Protein cIAP1 expression and Programmed Death - Ligand 1 expression. | Baseline
  The expression level of cIAP1 and the expression level of PD-L1 in biopsies will be measured by immunohistochemistry.
C. Correlation between the Inhibitor of Apoptosis Protein cIAP2 expression and Programmed Death - Ligand 1 expression. | Baseline
  The expression levels of cIAP2 and expression level of PD-L1 in biopsies will be measured by immunohistochemistry.
D. Correlation between the Inhibitor of Apoptosis Protein XIAP expression and lymphocytic tumour infiltration (LTI). | Baseline
  The expression level of XIAP and the level of lymphocytic tumour infiltration will be measured as % in biopsies.
D. Correlation between the Inhibitor of Apoptosis Protein cIAP1 expression and lymphocytic tumour infiltration (LTI). | Baseline
  The expression level of cIAP1 and the level of lymphocytic tumour infiltration will be measured as % in biopsies.
D. Correlation between the Inhibitor of Apoptosis Protein cIAP2 expression and lymphocytic tumour infiltration (LTI). | Baseline
  The expression level of cIAP2 and the level of lymphocytic tumour infiltration will be measured as % in biopsies.

OTHER OUTCOMES:
Age | Baseline
  Age will be recorded in years
Weight | Baseline
  Weight will be recorded in kilograms
Height | Baseline
  Height will be recorded in centimeters
Radiotherapy protocol | Baseline
  The patient's radiotherapy protocol will be recorded
Chemotherapy | Baseline
  Details of the patient's chemotherapy will be recorded (drugs and dosage)
Brachytherapy | Baseline
  Details of the patient's brachytherapy will be recorded (type of internal radiation and dosage)
Anatomopathology of cervical cancer: histology | Baseline
  The histology of the patient's cervical cancer will be recorded
Anatomopathology of cervical cancer: FIGO stage | Baseline
  The FIGO stage of the patient's cervical cancer will be recorded. FIGO staging ranges from Stage I= Confined to the uterine corpus and ovary to Stage IIB=Substantial lymphovascular space involvement of non-aggressive histological types.
Family and personal history | Baseline
  The patient's family and personal history will be recorded
Co-medications | Baseline
  Any other concommitant treatment will be recorded
Initial clinical features | Baseline
  The initial clinical features of the disease will be recorded
Lifestyle | Baseline
  The patient's lifestyle (marital status, children, hobbies, professional status) will be recorded
Follow-up | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  All details of follow-up of the patient's oncological pathology (response rate, date of progression, date of death) will be recorded.
Treatments received after progression | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Details of all treatments received after disease progression will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre TAYART de BORMS, Interne, Principal Investigator — Nîmes University Hospital; Cristina LEAHA, Dr., Principal Investigator — Institut Régional du Cancer de Montpellier, Service d'Anatomopathologie